CLINICAL TRIAL: NCT03580746
Title: Comparison of Ponseti Method Versus Older Treatments in Talipes Equinovarus Through Gait Analysis and Clinical Results
Status: Withdrawn | Type: Observational
Why Stopped: Resident working on this study left our department
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: UZLeuvenColette
Record Dates: First submitted 2014-09-23; First posted 2018-07-09 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Clubfoot
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Taping and posteromedial release: Children with clubfoots are treated by taping and posteromedial release
  Interventions: Procedure: Taping and posteromedial release
- Treatment by Ponseti: Children with clubfoots are treated by Ponseti
  Interventions: Procedure: Ponseti

INTERVENTIONS:
Procedure: Taping and posteromedial release
  Groups: Taping and posteromedial release
Procedure: Ponseti
  Groups: Treatment by Ponseti

SUMMARY:
There are many different treatments of congenital talipes equinovarus. At our institution, the investigators use the Ponseti method with manipulation and immobilization of the foot. In this study the investigators should like to demonstrate the better outcome in clinical results and in gait analysis of patients treated with the Ponseti method, compared to the 'older' methods of taping and posteromedial release.

DETAILED DESCRIPTION:
There are many different treatments of congenital talipes equinovarus. At our institution, the investigators use the Ponseti method with manipulation and immobilization of the foot. In this study the invistigators should like to demonstrate the better outcome in clinical results and in gait analysis of patients treated with the Ponseti method, compared to the 'older' methods of taping and posteromedial release. Trial objectives With this study the investigators would like to investigate whether clinical results and gait analysis in patients treated with Ponseti has better results compared to patients treated with the older methods.

ELIGIBILITY:
Inclusion Criteria:

* All patients with talipes equinovarus who have been treated at our institution

Exclusion Criteria:

* Patients with other disorders which may influence the clinical or gait analysis outcome

Ages: 2 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Retrospective study of children with club foots treated by two different options.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09 (Estimated); Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Clinical results | 1 year
  Different clinical results between the two groups using AOFAS (American Orthopaedic Foot and Ankle Society) score.

SECONDARY OUTCOMES:
Gait analysis | 1 year
  Differences in gait analysis between the two groups. While walking barefoot following parameters will be compared: ranges of motion occurring at each joint and each sub phase of stance

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leuven, Pellenberg, Vlaams-Brabant, Belgium